CLINICAL TRIAL: NCT01767090
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2 Study to Assess the Efficacy, Safety, and Dose-Response Relationship of ASP1707 in Subjects With Endometriosis Associated Pelvic Pain for 12 Weeks, Followed by a 12-Week Double-blind Extension Without Placebo Control, Including a 24-Week Open-Label Leuprorelin Acetate Treatment Group for Bone Mineral Density Assessment
Brief Title: A Study to Assess the Effectiveness and Safety of Different Doses of ASP1707 Compared to Placebo for Endometriosis Associated Pelvic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1707-CL-0011; 2012-002791-14 (EudraCT Number)
Record Dates: First submitted 2012-12-18; First posted 2013-01-14 (Estimated); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Endometriosis
Keywords: Phase 2; Double-blind; Pelvic pain; ASP1707; Placebo-controlled; Endometriosis
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — opigolix; Leuprolide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator): Applicable to first 12 week period (Part One); subjects in this arm will be randomized to one of the ASP1707 dose levels for the second 12 week period (Part Two)
  Interventions: Drug: Placebo
- ASP1707 lowest dose (Experimental): Subjects in this arm will be dosed with ASP1707 once daily for a total of 12 weeks (Part One) and continue taking the assigned dose for a further 12 weeks during the extension phase of the study (Part Two) for a total of 24 weeks
  Interventions: Drug: ASP1707
- ASP1707 low dose (Experimental): Subjects in this arm will be dosed with ASP1707 once daily for a total of 12 weeks (Part One) and continue taking the assigned dose for a further 12 weeks during the extension phase of the study (Part Two) for a total of 24 weeks
  Interventions: Drug: ASP1707
- ASP1707 medium dose (Experimental): Subjects in this arm will be dosed with ASP1707 once daily for a total of 12 weeks (Part One) and continue taking the assigned dose for a further 12 weeks during the extension phase of the study (Part Two) for a total of 24 weeks
  Interventions: Drug: ASP1707
- ASP1707 high dose (Experimental): Subjects in this arm will be dosed with ASP1707 once daily for a total of 12 weeks (Part One) and continue taking the assigned dose for a further 12 weeks during the extension phase of the study (Part Two) for a total of 24 weeks
  Interventions: Drug: ASP1707
- Leuprorelin acetate (Active Comparator): Subjects in this arm will be treated with leuprorelin acetate for a total of 24 weeks
  Interventions: Drug: Leuprorelin acetate

INTERVENTIONS:
Drug: ASP1707 — Oral
  Arms: ASP1707 high dose; ASP1707 low dose; ASP1707 lowest dose; ASP1707 medium dose
Drug: Placebo — Oral
  Arms: Placebo
Drug: Leuprorelin acetate — subcutaneous
  Other Names: Prostap® SR
  Arms: Leuprorelin acetate

SUMMARY:
The main objective for this study is to assess the efficacy and dose-response relationship of ASP1707 in reduction of endometriosis associated pelvic pain. The secondary objectives are to assess the safety, tolerability, Pharmacokinetics of ASP1707, dose response relationship of ASP1707 in reduction of E2 (Estradiol), 24-week efficacy of ASP1707 in reduction of endometriosis associated pain and 24-week safety and tolerability of ASP1707.

ELIGIBILITY:
Inclusion Criteria:

* Pre menopausal female adults with confirmed length and regular menstrual cycle
* Surgically diagnosed endometriosis
* Moderate to severe endometriosis related pain

Exclusion Criteria:

* Hormonal contraceptives or other drugs with effects on gynecological endocrinology
* Surgery for endometriosis within the 4 weeks prior to entry
* Uterine myoma
* Abnormal vaginal bleeding
* Hysterectomy or bilateral oophorectomy
* Pelvic infection
* Relevant abnormalities at gynecological exam at screening
* Disease with chronic abdominal pain of non-endometriosis origin
* Pituitary adenoma

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 912 (Actual)
Dates: Start 2012-12-04 (Actual); Primary Completion 2015-05-13 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the end of 12 weeks treatment of pain score for overall pelvic pain | Baseline & Week 12
Change from baseline to the end of 12 weeks treatment of pain score for dysmenorrhea | Baseline & Week 12
Change from baseline to the end of 12 weeks treatment of pain score for non-menstrual pelvic pain | Baseline & Week 12

SECONDARY OUTCOMES:
Change from baseline to the end of 24 weeks treatment of pain score for overall pelvic pain | Baseline & Week 24
Change from baseline to the end of 24 weeks treatment of pain score for dysmenorrhea | Baseline & Week 24
Change from baseline to the end of 24 weeks treatment of pain score for non-menstrual pelvic pain | Baseline & Week 24
Change from baseline to the end of treatment (EoT) of the dyspareunia score | Baseline, Week 12 & Week 24
Occurrence of response at the EoT for pain score for overall pelvic pain, dysmenorrhea, non-menstrual pelvic pain and dyspareunia | Week 12 & Week 24
Change from baseline to the EoT of the mean scores of the modified Biberoglu and Behrman (B&B) symptom and sign domains | Baseline, Week 12 & Week 24
Change from baseline to the EoT of the use of protocol defined rescue medication | Baseline, Week 12 & Week 24
Change from baseline to the EoT of the mean Pain Interference score of the Brief Pain Inventory | Baseline, Week 12 & Week 24
Patient Global Impression of Change (PGIC) at the End of Treatment | Week 12 & Week 24
Change from baseline to the EoT in the Endometriosis Health Profile (EHP)-5 score | Baseline, Week 12 & Week 24
Change from baseline to the EoT of the Female Sexual Function Index (FSFI) score (sexual well-being) | Baseline, Week 12 & Week 24
Change from baseline to the EoT of the Beck's Depression Inventory (BDI)-II score | Baseline, Week 12 & Week 24
Change from baseline to the EoT in the EuroQol (EQ-5D-5L) score | Baseline, Week 12 & Week 24
Safety and tolerability of ASP1707 measured by Adverse Events (AEs), bleeding patterns, Bone Mineral Density (BMD) | Up to Week 42
Pharmacodynamic profile of ASP1707 measured by Serum Estradiol (E2) levels | Up to Week 26
Pharmacokinetic profile of ASP1707 | Up to Week 24
  Both CL/F, V/F, AUCtau, Cmax, Ctrough

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (85):
- Belgium (5):
  - Site: 1006, Brussels
  - Site: 1002, Genk
  - Site: 1003, Ghent
  - Site: 1001, Leuven
  - Site: 1005, Liège
- Bulgaria (6):
  - Site: 1105, Plovdiv
  - Site: 1104, Sofia
  - Site: 1107, Sofia
  - Site: 1106, Sofia
  - Site: 1102, Sofia
  - Site: 1103, Stara Zagora
- Germany (5):
  - Site: 1390, Berlin
  - Site: 1304, Dresden
  - Site: 1302, Erlangen
  - Site: 1311, Karlsruhe
  - Site: 1306, Lübeck
- Hungary (7):
  - Site: 1422, Kecskemét, Bacs-Kiskun Megye
  - Site: 1401, Budapest
  - Site: 1407, Budapest
  - Site: 1408, Debrecen
  - Site: 1406, Pécs
  - Site: 1403, Szekszárd
  - Site: 1402, Székesfehérvár
- Japan (34):
  - Site: 2018, Aomori
  - Site: 2017, Chiba
  - Site: 2005, Fujisawa
  - Site: 2034, Hyōgo
  - Site: 2039, Hyōgo
  - Site: 2040, Hyōgo
  - Site: 2032, Kagoshima
  - Site: 2015, Kanagawa
  - Site: 2035, Kanagawa
  - Site: 2013, Kawagoe
  - Site: 2029, Kawasaki
  - Site: 2024, Kawasaki
  - Site: 2033, Kochi
  - Site: 2031, Kumamoto
  - Site: 2010, Kurashiki
  - Site: 2006, Kyoto
  - Site: 2036, Nagano
  - Site: 2037, Nagano
  - Site: 2038, Nagano
  - Site: 2002, Nagaoka
  - Site: 2007, Nagasaki
  - Site: 2011, Nara
  - Site: 2027, Sapporo
  - Site: 2001, Sapporo
  - Site: 2030, Sapporo
  - Site: 2004, Tokyo
  - Site: 2020, Tokyo
  - Site: 2014, Tokyo
  - Site: 2009, Tokyo
  - Site: 2003, Tokyo
  - Site: 2028, Tokyo
  - Site: 2025, Tokyo
  - Site: 2016, Tokyo
  - Site: 2012, Yokohama
- Poland (9):
  - Site: 1501, Bialystok
  - Site: 1505, Bialystok
  - Site: 1512, Gdansk
  - Site: 1504, Katowice
  - Site: 1508, Lublin
  - Site: 1507, Lublin
  - Site: 1502, Warsaw
  - Site: 1509, Warsaw
  - Site: 1525, Warzawa
- Romania (6):
  - Site: 1604, Brasov
  - Site: 1607, Bucaresti
  - Site: 1602, Bucharest
  - Site: 1601, Bucharest
  - Site: 1606, Bucharest
  - Site: 1603, Târgu Mureş
- Ukraine (9):
  - Site: 1701, Bucuresti
  - Site: 1702, Bucuresti
  - Site: 1705, Bucuresti
  - Site: 1707, Bucuresti
  - Site: 1713, Donetsk
  - Site: 1716, Donetsk
  - Site: 1708, Kyiv
  - Site: 1703, Targu Mures
  - Site: 1717, Zaporizhzhya
- United Kingdom (4):
  - Site: 1807, London
  - Site: 1804, Norwich
  - Site: 1808, Sheffield
  - Site: 1806, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] D'Hooghe T, Fukaya T, Osuga Y, Besuyen R, Lopez B, Holtkamp GM, Miyazaki K, Skillern L. Efficacy and safety of ASP1707 for endometriosis-associated pelvic pain: the phase II randomized controlled TERRA study. Hum Reprod. 2019 May 1;34(5):813-823. doi: 10.1093/humrep/dez028. PMID 31067329
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=305